CLINICAL TRIAL: NCT04220047
Title: Fuwai Hospital, Chinese Academy of Medical Science
Brief Title: Effects of Left Atrial Appendage Resection and Marshall Ligament Amputation on Clinical Outcome in Patients Undergoing Off-pump Coronary Artery Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-1304
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Stroke; Atrial Fibrillation
Keywords: off-pump coronary artery bypass; postoperative new-onset atrial fibrillation; left atrial appendage; Marshall ligament
MeSH Terms: conditions — Coronary Artery Disease; Stroke; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Atrial Appendage Resection (Experimental)
  Interventions: Procedure: Left Atrial Appendage Resection and Marshall Ligament Amputation
- off-pump coronary artery bypass (No Intervention)

INTERVENTIONS:
Procedure: Left Atrial Appendage Resection and Marshall Ligament Amputation — Left Atrial Appendage Resection and Marshall Ligament Amputation during the cardiac surgery
  Arms: Left Atrial Appendage Resection

SUMMARY:
Surgical occlusion of the left atrial appendage (LAAO) is sometimes performed during the cardiac surgery to reduce long-term risk of stroke.A previous study found that LAAO may be associated with increased risk of postoperative atrial fibrillation.New-onset atrial fibrillation (NOAF) after coronary artery bypass graft is related to an increased short-term and long term risk of stroke and mortality.Marshall ligament amputation may reduce the occurence of atrial fibrillation. However, little is known whether this approach is justified during the coronary artery bypass graft.Therefore, this study aimed to investigate whether LAAO and Marshall ligament amputation during off-pump coronary artery bypass was associated with reduced risks of postoperative new-onset atrial fibrillation and stroke.

ELIGIBILITY:
Inclusion Criteria:

* isolated first off-pump coronary artery bypass

Exclusion Criteria:

* Preoperative atrial fibrillation or a history of atrial fibrillation;
* Concurrent cardiac or non-cardiac surgery
* Intraoperative convert to bypass bypass surgery
* Emergency surgery
* History of previous cardiac surgery
* Severe organ dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative new-onset atrial fibrillation | 7 days
  Postoperative atrial fibrillation (POAF), defined as new-onset atrial fibrillation (AF) in the immediate period after surgery, is the most important type of secondary AF.

SECONDARY OUTCOMES:
stroke | 1 months,3 months, 1years, 3years, 5years.
  Stroke is caused by a disruption in the flow of blood to part of the brain either because of occlusion of a blood vessel in the case of acute ischemic stroke （AIS） or the rupture of a blood vessel causing bleeding in or around the brain： intracerebral hemorrhage （ICH）or subarachnoid hemorrhage （SAH）。

CONTACTS AND LOCATIONS:
Overall Officials: Hansong Sun, doctor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, China